CLINICAL TRIAL: NCT05890352
Title: Randomized Phase II Study of the Addition of Targeted Therapeutic Agents to Tafasitamab-Based Therapy in Non-Transplant-Eligible Patients With Relapsed/Refractory Large B-Cell Lymphoma
Brief Title: Study Adding Drugs to Usual Treatment for Large B-Cell Lymphoma That Returned or Did Not Respond to Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); BeiGene (Industry); Ipsen (Industry); Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: S2207; NCI-2023-02518 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2207 (Other: SWOG); S2207 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Grade 3b Follicular Lymphoma; High Grade B-Cell Lymphoma; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; Recurrent Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Transformed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Specimen Handling; Lenalidomide; Magnetic Resonance Spectroscopy; tafasitamab; Immunoglobulins; Disulfides; tazemetostat; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part I, Arm I (tafasitamab, lenalidomide, tazemetostat) (Experimental): Patients receive tafasitamab IV, lenalidomide PO, and tazemetostat PO on study. Patients also undergo PET/CT and CT or MRI scans throughout the trial. Patients also have the option to undergo collection of blood samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Biological: Tafasitamab; Drug: Tazemetostat
- Part I, Arm III (tafasitamab, lenalidomide, zanubrutinib) (Experimental): Patients receive tafasitamab IV, lenalidomide PO, and zanubrutinib PO on study. Patients also undergo PET/CT and CT or MRI scans throughout the trial. Patients also have the option to undergo collection of blood samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Tafasitamab; Drug: Zanubrutinib
- Part II, Arm I (tafasitamab, lenalidomide, tazemetostat) (Experimental): Patients receive tafasitamab IV, lenalidomide PO, and tazemetostat PO on study. Patients also undergo PET/CT and CT or MRI scans throughout the trial. Patients also have the option to undergo collection of blood samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Tafasitamab; Drug: Tazemetostat
- Part II, Arm II (tafasitamab, lenalidomide) (Active Comparator): Patients receive tafasitamab IV and lenalidomide PO on study. Patients also undergo PET/CT and CT or MRI scans throughout the trial. Patients also have the option to undergo collection of blood samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Tafasitamab
- Part II, Arm III (tafasitamab, lenalidomide, zanubrutinib) (Experimental): Patients receive tafasitamab IV, lenalidomide PO, and zanubrutinib PO on study. Patients also undergo PET/CT and CT or MRI scans throughout the trial. Patients also have the option to undergo collection of blood samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Tafasitamab; Drug: Zanubrutinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo optional collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT and CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
  Arms: Part I, Arm III (tafasitamab, lenalidomide, zanubrutinib); Part II, Arm I (tafasitamab, lenalidomide, tazemetostat); Part II, Arm II (tafasitamab, lenalidomide); Part II, Arm III (tafasitamab, lenalidomide, zanubrutinib)
Biological: Tafasitamab — Given IV
  Other Names: Immunoglobulin, Anti-(Human Cd19 Antigen) (Human-mus musculus Monoclonal MOR00208 Heavy Chain), Disulfide with Human-mus musculus Monoclonal MOR00208 .Kappa.-chain, Dimer; Monjuvi; MOR-00208; MOR00208; MOR208; Tafasitamab-cxix; XmAb5574
Drug: Tazemetostat — Given PO
  Other Names: E7438; EPZ-6438; EPZ6438
  Arms: Part I, Arm I (tafasitamab, lenalidomide, tazemetostat); Part II, Arm I (tafasitamab, lenalidomide, tazemetostat)
Drug: Zanubrutinib — Given PO
  Other Names: BGB-3111; Brukinsa; BTK-InhB
  Arms: Part I, Arm III (tafasitamab, lenalidomide, zanubrutinib); Part II, Arm III (tafasitamab, lenalidomide, zanubrutinib)

SUMMARY:
This phase 2 trial studies the side effects and best dose of tazemetostat and zanubrutinib in combination with tafasitamab and lenalidomide, and to see how well these combinations work in treating patients with large B-cell lymphoma that returned or did not respond to earlier treatment. Tazemetostat is in a class of medications called EZH2 inhibitors. It helps to stop the spread of cancer cells. Zanubrutinib is in a class of medications called kinase inhibitors. It works by blocking the action of the abnormal protein that signals cancer cells to multiply. This helps stop the spread of cancer cells. tafasitamab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Lenalidomide is in a class of medications called immunomodulatory agents. It works by helping the bone marrow to produce normal blood cells and by killing abnormal cells in the bone marrow. The addition of tazemetostat or zanubrutinib to tafasitamab and lenalidomide may be able to shrink the cancer or extend the time without cancer symptoms coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose of tafasitamab + lenalidomide + tazemetostat AND of tafasitamab + lenalidomide + zanubrutinib. (Safety Run-in) II. To compare progression-free survival (PFS) of patients with relapsed/refractory large B-cell lymphoma (R/R LBCL) treated with tafasitamab + lenalidomide + tazemetostat vs control (tafasitamab + lenalidomide) AND treated with tafasitamab + lenalidomide + zanubrutinib versus (vs) control. (Randomized Phase II Study)

SECONDARY OBJECTIVES:

I. To estimate the hazard ratio for PFS for control vs. tafasitamab + lenalidomide + tazemetostat in germinal center B-cell (GCB) and non-GCB (activated B-cell [ABC]/unclassified) subsets.

II. To estimate the hazard ratio for PFS for control vs. tafasitamab + lenalidomide + zanubrutinib in GCB and non-GCB (ABC/unclassified) subsets.

III. To estimate progression-free survival (PFS), overall response rate (ORR), complete response rate (CR), partial response rate (PR), duration of response (DOR), event-free survival (EFS), overall survival (OS), in GCB and non-GCB LBCL for each treatment.

IV. To evaluate adverse events within each treatment arm.

OTHER OBJECTIVES:

I. To explore PFS within subgroups defined by molecular profile (e.g., MCD, BN2, N1 and EZB) and genetic subtypes.

II. To explore PFS in the tafasitamab-lenalidomide control arm vs that in matched historical control from L-MIND and realMIND studies.

III. To assess frailty (Cumulative Illness Rating Scale [CIRS] and Timed Get Up and Go [TUG]) and its correlation with outcome.

PRIMARY PATIENT-REPORTED OUTCOMES OBJECTIVE:

I. To compare patient-reported lymphoma-specific symptoms as measured by the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) Trial Outcome Index sub-scale at 3 months after randomization between the control arm and each experimental arm (Arm 1 versus Arm 2 and Arm 3 versus Arm 2).

SECONDARY PATIENT-REPORTED OUTCOMES OBJECTIVE:

I. To compare participant-reported toxicity (treatment side effect) symptoms using selected Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) items between experimental vs control arms.

EXPLORATORY PATIENT-REPORTED OUTCOMES OBJECTIVES:

I. To compare patient-reported quality of life using the FACT-General (G) subscale score and the FACT-Lym total score at 3 months after randomization between the control arm and each experimental arm.

II. To compare quality of life over time between treatment arms from baseline to 12 months after randomization as measured by the FACT-Lym trial outcome index (TOI), FACT-G, and FACT-Lym total score using longitudinal analysis.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE: This is a dose-escalation study of tazemetostat and zanubrutinib.

PART I (SAFETY RUN-IN): Patients are assigned to 1 of 2 arms per treating investigator's choice.

ARM I: Patients receive tafasitamab intravenously (IV), lenalidomide orally (PO), and tazemetostat PO on study. Patients also undergo positron emission tomography/computed tomography (PET/CT) and CT or magnetic resonance imaging (MRI) scans throughout the trial. Patients also have the option to undergo collection of blood samples during screening and on study.

ARM III: Patients receive tafasitamab IV, lenalidomide PO, and zanubrutinib PO on study. Patients also undergo PET/CT and CT or MRI scans throughout the trial. Patients also have the option to undergo collection of blood samples during screening and on study.

PART II: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive tafasitamab IV, lenalidomide PO, and tazemetostat PO on study. Patients also undergo PET/CT and CT or MRI scans throughout the trial. Patients also have the option to undergo collection of blood samples during screening and on study.

ARM II: Patients receive tafasitamab IV and lenalidomide PO on study. Patients also undergo PET/CT and CT or MRI scans throughout the trial. Patients also have the option to undergo collection of blood samples during screening and on study.

ARM III: Patients receive tafasitamab IV, lenalidomide PO, and zanubrutinib PO on study. Patients also undergo PET/CT and CT or MRI scans throughout the trial. Patients also have the option to undergo collection of blood samples during screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have:

  * Histologically confirmed relapsed/refractory LBCL as outlined by the World Health Organization (WHO) guidelines
  * Follicular lymphoma, grade 3B
  * Transformed lymphoma
  * High grade B-cell lymphoma with or without MYC, BCL2 and/or BCL6 rearrangements
* Participants must have staging imaging performed within 28 days prior to registration, as follows. Positron emission tomography (PET)-computed tomography (CT) baseline scans are strongly preferred; diagnostic quality magnetic resonance imaging (MRI), contrast-enhanced CT, or contrast-enhanced MRI scans are also acceptable if PET-CT is not feasible at baseline. Note: PET-CT will be required at end of treatment (EOT) and progression for response assessment. All measurable lesions (longest diameter >= 1.5 cm) must be assessed within 28 days prior to registration. Tests to assess non-measurable disease must be performed within 28 days prior to registration. All disease must be documented on the Baseline Tumor Assessment Form.
* Participants must have cell of origin (COO) determination of germinal center (GC)(GCB or non-GC GCB) of LBCL based on Hans immunohistochemistry algorithm (CD10, BCL6, MUM1) as noted on pathology report.
* Participants must have had 1-5 prior systemic treatment regimens including one systemic multiagent regimen for aggressive lymphoma
* Participants who have received prior systemic therapy must have completed their last treatment prior to registration. Participants must have recovered from previous therapy
* Steroid use for the control of non-Hodgkin lymphoma symptoms is allowable, but must be discontinued prior to Cycle 1, Day 1
* Participant must be >= 18 years old
* Participant must have Zubrod Performance Status of 0-3
* Participant must have a complete medical history and physical exam within 28 days prior to registration
* Absolute neutrophil count >= 1.0 x 10^3/uL (within 28 days prior to registration)

  * If there is documented lymphomatous involvement of the bone marrow as assessed by bone marrow biopsy within 90 days prior to registration, participants must have: Absolute neutrophil count (ANC) >= 0.75 x 10^3/uL
* Platelets >= 75 x 10^3/uL (within 28 days prior to registration)

  * If there is documented lymphomatous involvement of the bone marrow as assessed by bone marrow biopsy within 90 days prior to registration, participants must have: Platelets >= 50 x 10^3/uL
* Aspartate aminotransferase (AST) =< 3 x institutional upper limit of normal (IULN), alanine aminotransferase (ALT) =< 3 x IULN (within 28 days prior to registration) unless due to Gilbert's disease, hemolysis, or lymphomatous involvement of liver.

  * Participants with lymphomatous involvement of the liver must have AST =< 5 x IULN, ALT =< 5 x IULN
* Total bilirubin =< 1.5 x IULN (within 28 days prior to registration) unless due to Gilbert's disease, hemolysis, or lymphomatous involvement of liver.

  * Participants with lymphomatous involvement of the liver must have total bilirubin =< 5 x IULN
* Participants must have a calculated creatinine clearance >= 30 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to registration
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Participants must have recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia
* Participants with known human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at randomization and have undetectable viral load test on the most recent test results obtained within 6 months prior to registration
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on the most recent test results obtained within the last year and received suppressive therapy
* Participants with a history of hepatitis C virus (HCV) infection must have an undetectable viral load. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 28 days prior to registration
* Participants must be able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption, such as malabsorption syndrome or major resection of the stomach or bowels
* Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System
* Participants who can complete the FACT-Lym and PRO-CTCAE forms in English or Spanish must agree to participate in the patient-reported outcome study
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines.

  * For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and central institutional review board (CIRB) regulations.

Exclusion Criteria:

* Participants must not have active lymphomatous involvement of the central nervous system (CNS) because the treatments used in this study are not effective to sufficiently penetrate the blood brain barrier
* Participants must not have known abnormalities associated with myelodysplastic syndrome (MDS) (e.g., del 5q, chr 7 abn) and myeloproliferative neoplasms (MPN) (e.g., JAK2 V617F) observed in cytogenetic testing and deoxyribonucleic acid (DNA) sequencing. Testing is not required for eligibility determination
* Participants must not have a known prior history of T-cell lymphoblastic lymphoma (T-LBL)/T-cell acute leukemia (T-ALL). Testing is not required for eligibility determination
* Participants must not be a candidate based on investigator assessment to receive autologous stem cell transplant (ASCT) or must have declined ASCT. Participants who had disease progression after stem cell transplant or cellular therapy (such as chimeric antigen receptor (CAR) T-cell) are eligible
* Participants must not have received prior treatment with tafasitamab and/or lenalidomide
* Participants must not have had prior BTK inhibitor or tazemetostat
* Participants must not have any known allergy or reaction to any component of tafasitamab, lenalidomide, tazemetostat or zanubrutinib
* Participants must not be receiving direct vitamin K inhibitors or strong or moderate CYP3A inhibitors or inducers at the date of registration

  * Notes: Because the list of these agents is constantly changing, it is important to regularly consult a frequently updated medical reference
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not be pregnant or nursing and must follow the guidelines according to the lenalidomide Risk Evaluation and Mitigation Strategies (REMS) program. The effects of tazemetostat, zanubrutinib, lenalidomide and tafasitamab, and the combination of these drugs have not been studied on the developing human fetus are the effects are unknown. Individuals who are of reproductive potential must have agreed to use a highly effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential". In addition to routine contraceptive methods, "acceptable contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization to date of first observation of progressive disease according to the 2014 Lugano classification, or death due to any cause, assessed up to 3 years
  Will be compared between participants randomized to control Arm 2 (tafasitamab + lenalidomide) versus (vs) experimental Arm 1 (tafasitamab + lenalidomide + tazemetostat), AND control Arm 2 vs experimental Arm 3 (tafasitamab + lenalidomide + zanubrutinib), respectively.
Trial Outcome Index (TOI) score from the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) (Patient Reported Outcome [PRO] Study) | Baseline up to 3 months after randomization
  Will compare the trial outcome index (TOI) score between each experimental arm (Arm 1 and Arm 3) to the control arm (Arm 2). The TOI score is composed of the Physical Well-Being, Functional Well-Being, and lymphoma-specific subscale scores. The scores range from 0-116, with higher scores indicating a higher quality of life.

SECONDARY OUTCOMES:
Hazard ratio for PFS in the germinal center B-cell (GCB) subgroup | Up to 3 years
  Will calculate the 80% confidence interval (CI) for the Cox regression time-to-event estimate of the hazard ratio associated with addition of tazemetostat to tafasitamab+lenalidomide combination (Arm 2 vs Arm 1) in the GCB subgroup. If the confidence interval excludes 1, then 80% CI will be calculated for the non-GCB group.
Hazard ratio for PFS in the non-GCB subgroup | Up to 3 years
  Will calculate the 80% CI for the hazard ratio associated with addition of zanubrutinib to tafasitamab+lenalidomide combination (Arm 2 vs Arm 3) in the non-GCB subgroup. If the confidence interval excludes 1, then 80% CI will be calculated for the GCB group.
PFS | From date of randomization to date of first observation of progressive disease according to the 2014 Lugano classification, or death due to any cause, assessed up to 3 years
  Will estimate in GCB and non-GCB large B-cell lymphoma (LBCL) for each treatment. Will be estimated using the method of Kaplan-Meier and 80% confidence interval will be calculated.
Overall response rate (ORR) | Up to 3 years
  Will estimate in GCB and non-GCB LBCL for each treatment. Will be estimated using the method of Kaplan-Meier and 80% confidence interval will be calculated.
Complete response (CR) rate | Up to 3 years
  Will estimate in GCB and non-GCB LBCL for each treatment. Will be estimated using the method of Kaplan-Meier and 80% confidence interval will be calculated.
Partial response (PR) rate | Up to 3 years
  Will estimate in GCB and non-GCB LBCL for each treatment. Will be estimated using the method of Kaplan-Meier and 80% confidence interval will be calculated.
Duration of response (DOR) | From date of first documentation of response to treatment (CR, PR) to date of first documentation of progression, or death due to any cause among patients who achieve a response (CR or PR), assessed up to 3 years
  Will estimate in GCB and non-GCB LBCL for each treatment. Will be estimated using the method of Kaplan-Meier and 80% confidence interval will be calculated.
Event free survival (EFS) | From date of randomization to date of first occurrence of EFS event, assessed up to 3 years
  Will estimate in GCB and non-GCB LBCL for each treatment. Will be estimated using the method of Kaplan-Meier and 80% confidence interval will be calculated.
Overall survival (OS) | From date of randomization to date of death due to any cause, assessed up to 3 years
  Will estimate in GCB and non-GCB LBCL for each treatment. Will be estimated using the method of Kaplan-Meier and 80% confidence interval will be calculated.
Incidence of adverse events | Up to 3 years
  Will be evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5. Eligible participants receiving at least one dose of drug will be included in the assessment of adverse events by treatment arms. The maximum Grade for each toxicity will be recorded for each participant, and frequency tables will be reviewed to determine toxicity patterns. With 60 eligible participants in each arm, any toxicity occurring with at least 5% probability is likely to be seen at least once (95% chance). Toxicity rates in each arm can be estimated to within at least +/- 13% with 95% confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Amengual, Principal Investigator — SWOG Cancer Research Network
Locations (104):
- United States (104):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Seacliff, Huntington Beach, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - City of Hope Newport Beach, Newport Beach, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin